CLINICAL TRIAL: NCT00588913
Title: Phase I/II Study of Adoptive Immunotherapy Comprising Pyrophosphomonoester Antigen-stimulated T Cells, IL-2, and Nitrogen-containing Bisphosphonates in Patients With Stage IV Renal Cell Carcinoma
Brief Title: Adoptive Immunotherapy, Aldesleukin, and Zoledronate in Treating Patients With Stage IV Kidney Cancer and Lung Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tokyo Women's Medical University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: TRIC-CTR-GU-05-01; CDR0000581156 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2007-12-20; First posted 2008-01-09 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2009-08

CONDITIONS: Kidney Cancer; Metastatic Cancer
Keywords: recurrent renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma; lung metastases
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — aldesleukin; Zoledronic Acid

INTERVENTIONS:
Biological: aldesleukin
Biological: therapeutic autologous lymphocytes
Drug: zoledronic acid

SUMMARY:
RATIONALE: Cellular adoptive immunotherapy uses a person's white blood cells that are treated in the laboratory to stimulate the immune system in different ways and stop tumor cells from growing. Aldesleukin may help the laboratory-treated white blood cells stay in the body longer. Drugs used in chemotherapy, such as zoledronic acid, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving cellular adoptive immunotherapy together with interleukin-2 and zoledronic acid may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects of giving cellular adoptive immunotherapy together with aldesleukin and zoledronic acid and to see how well it works in treating patients with stage IV kidney cancer and lung metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of adoptive immunotherapy comprising 2-methyl-3-butenyl-1-pyrophosphate-stimulated gamma delta (gd) T cells, zoledronate, and IL-2 after nephrectomy, especially with regard to the incidence and frequency of adverse events.
* Determine the duration of in vivo persistence of the transferred gd T cells in patients.
* Determine the doubling time of tumor growth before and after adoptive immunotherapy.
* Determine the tumor-size reducing effect of adoptive immunotherapy based on the Best Overall Response Chart.

OUTLINE: Patients undergo leukapheresis for the harvest of peripheral blood mononuclear cells (PBMCs). PBMCs are stimulated with 2-methyl-3-butenyl-1-pyrophosphate and aldesleukin for 11 days. Patients then receive the expanded Gamma Delta T cells, aldesleukin, and zoledronic acid once a month for 6 months.

After completion of study treatment, patients are followed for up to 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed renal carcinoma

  * Stage IV disease with lung metastases
* Bidimensionally measurable lung metastases by CT scan
* Meets 1 or more of the following criteria:

  * No change in disease status or progressive disease after prior aldesleukin administration for 3 months or more
  * Lung metastases after treatment with prior nephrectomy
* Patients with clear cell renal carcinoma must have undergone nephrectomy prior to study entry

  * Patients with progression of metastatic lung cancer after nephrectomy also must have received interferon alfa for 3 months or more (prior to study entry)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Life expectancy > 6 months
* Leukocyte count ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum bilirubin ≤ 1.5 mg/dL
* AST/ALT ≤ 2.5 times normal
* Serum creatinine ≤ 1.7 mg/dL
* LDH ≤ 1.5 times normal
* Not pregnant nor nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection with hepatitis virus or HIV
* No poorly controlled heart failure or arrhythmia
* No hypercalcemia that require medication
* No C-reactive protein with an infectious disease that requires medication

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy, radiation therapy, or biologic therapy
* No prior bone marrow transplantation or organ transplantation
* No concurrent steroid therapy
* No concurrent antidepressant therapy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-03 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events based on NCI-CTCAE version 3.0
Proportion of gd T-cells in peripheral blood

SECONDARY OUTCOMES:
Secondary doubling time of tumor growth
Overall response

CONTACTS AND LOCATIONS:
Overall Officials: Hirohito Kobayashi, Study Chair — Tokyo Women's Medical University
Locations (2):
- Japan (2):
  - Kyoto University Hospital, Kyoto, Kyoto
  - Tokyo Women's Medical University, Tokyo, Tokyo